CLINICAL TRIAL: NCT06365944
Title: Concussion in French Non-professional Handball League : Efficiency of a Concussion Protocol, the White Card Process
Acronym: PRECCOCE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/73
Record Dates: First submitted 2024-03-29; First posted 2024-04-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Brain Concussion; Cerebral Concussion
Keywords: Sport-related Concussion; Handball; Epidemiology
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sport related concussion is a major issue for many contact sports, such as Rugby, Football, Hockey and Handball. As a response, some federations like World Rugby set up a concussion protocol, that starts with the referee having the responsibility to issue a blue card when suspecting a concussed player and thus have him off the field for medical examination. The French handball federation (FFHB) as well as its concussion protocol called "Protocole carton blanc", in this study we aim to describe the efficiency of this protocol.

DETAILED DESCRIPTION:
Sport related concussion is a major issue for many contact sports, such as Rugby, Football, Hockey and Handball. The short, medium and long-term issues of such impact are still debated but some studies have pointed the fact that acute concussion, repetitive concussions, and even "sub-concussive" impacts could major the risk of developing brain diseases and cognitive impairments. As a response, some federations like World Rugby set up a concussion protocol, that starts with the referee having the responsibility to issue a blue card when suspecting a concussed player and thus have him off the field for medical examination. The French handball federation (FFHB) as well as its concussion protocol called "Protocole carton blanc", in this study we aim to describe the efficiency of this protocol.

This study will be an epidemiological descriptive and prospective study with a brief questionnaire sent off to any player, above 18 years old, male or female, that had receive a white card during an official match in the French amateur Handball league along two regular season. The results will bring details on how concussion occurs on field and how this protocol is efficient to bring the player to consult a health professional.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 18 years old
* Who had received a white card during an official game
* having an email address registered in the FFHB register

Exclusion Criteria:

* Any refusal to participate
* Inability to respond

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is descriptive, prospective, with a questionnaire sent off to any player, above 18 years old, male or female, that had receive a white card during an official match in the French amateur Handball league along two regular season.During an official game, if the referee issues a white card, the player is then contacted by the French Handball Federation (FFHB) via an email in a day.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Proportion, as a percentage, of participant declaring no medical care while being estimated at risk of having a concussion (assessed by answers to the questionnaire) | Day 0
  Risk of concussion estimated by questionnaire collecting the following informations :
  - Sport Concussion Assessment Tool 6 (SCAT6)'s 22 symptoms, each symptoms is scales from 0 to 6, 6 being the highest intensity of the symptom.
  Having > 1 in at least two different symptoms is considered at risk of having a concussion

CONTACTS AND LOCATIONS:
Overall Officials: Helene CASSOUDESALLE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France